CLINICAL TRIAL: NCT00806390
Title: GCC0766: Prevention of Anthracycline or Trastuzumab Induced Cardiomyopathy by Metoprolol
Brief Title: Prevention of Anthracycline or Trastuzumab Induced Cardiomyopathy by Metoprolol
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Stephen Gottlieb, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HP-00040965
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Results first posted 2014-07-22 (Estimated); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Cardiomyopathy
Keywords: ejection fraction; anthracyclines; beta-adrenergic blockade; Patients receiving anthracyclines
MeSH Terms: conditions — Cardiomyopathies | interventions — Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metoprolol (Active Comparator): Receiving metoprolol
  Interventions: Drug: Metoprolol
- Control (No Intervention): Not receiving metoprolol

INTERVENTIONS:
Drug: Metoprolol — Metroprolol tartrate titrated up
  Arms: Metoprolol

SUMMARY:
The primary objective of this study is to investigate whether giving prophylactic metoprolol prior to and during anthracycline or trastuzumab therapy will decrease the incidence of anthracycline-induced cardiomyopathy. Patients are randomized to receive metoprolol or no treatment prior to anthracycline or trastuzumab treatment. The ejection fraction, as measured by nuclear ventriculography is measured before and after treatment.

DETAILED DESCRIPTION:
This is a randomized, controlled exploration. Consent will be obtained from patients receiving care for cancer with anthracycline or trastuzumab at the University Of Maryland Greenebaum Cancer Center prior to initiation of anthracycline or trastuzumab treatment during the initial oncology visit.

Patients will be evaluated in the initial consultation in the oncology clinic during which time consent will be obtained, and any patient with bradycardia (HR less than 50) or other contraindication will be excluded from the study. The patients will be randomly assigned to metoprolol vs. control groups during this initial visit. Individuals in the control group will not receive any study drug where as those in the metoprolol group will be given prophylactic metoprolol prior to initiation of anthracycline or trastuzumab treatment. Metoprolol tartrate will be provided to each patient randomized to the metoprolol group.

Also at the time of the initial consultation, a baseline MUGA will be obtained for evaluation of left ventricular ejection fraction. Additionally, a post-treatment MUGA will be obtained after the final course of chemotherapy. Lastly, also at the initial visit, one vial of blood will be obtained from each patient to test for genetic polymorphisms, as described in the background section, which may contribute to the response to beta blockade in the prevention of anthracycline or trastuzumab induced cardiomyopathy.

Each participant in the metoprolol group will be started on 25 mg of metoprolol tartrate twice a day prior to initiation of the anthracycline or trastuzumab. After one week, this dose will be increased to 50 mg twice daily, if tolerated. Prior to increasing the dose, the patients will be seen in the cardiology research clinic by the study doctor and evaluated for side effects. After another week the dose will again be increased to 100 mg twice daily. The dose can be decreased at any time if side effects occur such as bradycardia with HR less than 50 or hypotension with SBP less than 90. The beta blocker will be held for two days prior to the post-treatment MUGA so as not to acutely affect heart rate, as a decrease in heart rate would be expected to increase EF14. Abrupt cessation of metoprolol tartrate will not lead to withdrawal of beta-blockade. This study will end with the post-treatment MUGA. The primary end point of this study will be the change in EF before and after anthracycline or trastuzumab treatment. A pill diary will be maintained to document compliance of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have confirmed malignancy for which standard regimens of anthracyclines or trastuzumab are being offered as treatment at the University of Maryland Greenebaum Cancer Center. Patients must either receive 4 cycles of anthracycline for a total dose of 240 mg/m2 or six cycles of TAC for a total dose of 300 mg/m2 or trastuzumab.
2. Age > 18 years
3. Ability to understand and willingness to sign a written informed consent document.
4. Women of childbearing potential may participate in this study only if they have a negative pregnancy test and agree not to become pregnant during the study. Woman of childbearing potential must use an effective method of birth control such as hormonal contraceptives (oral and implant) condoms, diaphragms, spermicidal foam or jelly, surgical (hysterectomy or tubal ligation) or intrauterine device.

Exclusion Criteria:

1. Patients who have established dilated or restrictive cardiomyopathy with EF < 40 %.
2. Patients with severe mitral or aortic valve disease (valve area <1cm squared).
3. Patients who have any contraindication to metoprolol, in particular bradycardia with HR < 50, or severe reactive pulmonary disease such as asthma. Patients who take mibefradil or psychiatric drugs (such as phenothiazines including chlorpromazine and thioridazine) will also be excluded from the study as they have serious interactions with beta-blockers
4. Patients who have untreated thyroid function disorder.
5. Pregnant and nursing women are excluded from this study because of potential risk for adverse events to the fetus.
6. Patients with any impediment to swallowing tablets would be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-07; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen S Gottlieb, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metoprolol | Control
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoprolol | Control | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (11) | 47 (8) | 49 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Ejection Fraction by MUGA
Description: Because of the inability to enroll an adequate number of patients, (only 15 out of a planned 50) no data analysis was collected or performed.
Time Frame: Pre and post anthracycline treatment
Population: This study was unable to enroll a sufficient number of patients to permit analysis (only 15 patients enrolled)
Arm/Group | Metoprolol | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Metoprolol | Control
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No